CLINICAL TRIAL: NCT02734251
Title: Effects of Magnolia and Phellodendron (Magnolia Officinalis and Phellodendron Amurense) Bark Extracts on Anxiety, Cognitive Performance, and Mood Tested After Induced Stress
Brief Title: Effect of Relora Supplement on Anxiety, Cognitive Performance & Mood Tested After Induced Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InterHealth Nutraceuticals, Inc. (Industry)
Collaborators: MB Clinical Research, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MC-1514
Record Dates: First submitted 2016-04-05; First posted 2016-04-12 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Mood (Psychological Function)
Keywords: Healthy mood; Stress management; Relora; Healthy subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Dietary Supplement: Placebo
  Interventions: Dietary Supplement: Placebo
- Relora (Experimental): Dietary Supplement: Relora, 750 mg/day
  Interventions: Dietary Supplement: Relora

INTERVENTIONS:
Dietary Supplement: Relora — 750 mg/day
  Arms: Relora
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The present randomized, double-blind, placebo-controlled crossover trial aims to evaluate the effects of Relora supplementation on responses to induced stress produced by a combination of cognitive and physiologic stressors in healthy men and women. The effects of the supplement, compared with a placebo, will be evaluated using measures to assess anxiety [State-Trait Anxiety Inventory-Part 1 (STAI-Part 1), mood [Bond-Lader Visual Analog Scale (VAS)], hypothalamic-pituitary-adrenal axis activation (salivary cortisol) and cognitive function (cognitive flexibility, reaction time, processing speed, attention, sustained attention, working memory, and executive function). Testing will be completed at the beginning and end of 7-d supplementation periods with the active and placebo products to assess both the acute effects and the "acute-on-chronic" effects following one week of daily use.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female, 21-59 years of age, inclusive.
2. Subject is judged by the Investigator to be in general good health on the basis of medical history and screening laboratory tests.
3. Subject has a BMI of 18.50-29.99 kg/m2, inclusive, at visit 1 (day -6).
4. Subject is a non-user of nicotine products for 6 months prior to visit 1 (day -6).
5. Subject is willing to maintain a habitual diet and physical activity patterns throughout the study period.
6. Subject is willing and able to attend the screening visit and 4 test visits lasting up to ~4 h each (visits 2 through 5; days 1 and 7 of Period I and Period II, respectively).
7. Subject is able to maintain immersion of non-dominant hand, including the forearm, into ice water (0-4°C) for ≥30 seconds during the CPT at visit 1 (day -6).
8. Subject is willing to refrain from alcohol for 12 h prior to each test visit (visits 2 through 5; days 1 and 7 of Periods I and II, respectively) and to limit alcohol consumption to no more than one serving of alcohol (1 drink = 12 oz beer, 5 oz wine, or 1.5 oz hard liquor) the 24 h prior to each test visit (visits 2, 3, 4, and 5; days 1 and 7 of Period I and Period II, respectively).
9. Subject is willing to limit caffeine-containing beverages/foods/products consumed at the breakfast meal on all test visit days (visits 2, 3, 4, and 5; days 1 and 7 of Period I and Period II, respectively) to no more than 1 serving (150 mg) ≥2 h prior to each test visit.
10. Subject is willing to consume a hearty breakfast on a daily basis throughout the study period with replication of the timing and quantities of food and beverages consumed at the visit 2 (day 1) breakfast meal on the morning of each subsequent test visit (visits 3 through 5; day 7 of Period I and days 1 and 7 of Period II).
11. Subject is willing to replicate the timing and dose of any necessary morning medications and/or supplements taken prior to coming to clinic on visit 2 (day 1) at each subsequent test visit (visits 3 through 5; day 7 of Period I and days 1 and 7 of Period II).
12. Subject is willing and able to comfortably abstain from caffeine throughout the duration of all test visits (~5 h; visits 2, 3, 4, and 5; days 1 and 7 of Period I and Period II, respectively).
13. Subject understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator and is willing to complete study procedures.

Exclusion Criteria:

1. Subject has a history or presence of clinically important cardiac, renal, hepatic, endocrine (including Type 1 and Type 2 diabetes mellitus), pulmonary, biliary, pancreatic, or neurologic disorders.
2. Subject has a history of diagnosed generalized anxiety, and/or other major psychiatric disorder(s), other than diagnosed depression.
3. Subject has a history of diagnosed depression in the 2 years prior to visit 1 (day -6) and/or a score of 17 or higher on the Beck Depression Scale.
4. Subject has an abnormal comprehensive metabolic panel and/or complete blood count test result of clinical significance. A reflex HbA1C may be assessed on subjects with a blood glucose ≥126 mg/dL to determine glycemic status, at discretion of Investigator.
5. Subject tests positive for any of the substances included in urine drug screen (i.e., cocaine, tetrahyrdocannabinol, opiates, amphetamines, methamphetamines, phencyclidines, benzodiazepines, barbiturates, methadone, oxycodone, methylenedioxymethamphetamine, and propoxyphene).
6. Subject is unable to understand and/or perform required tests based on the practice test results.
7. Subject has a history of unconventional sleep patterns (e.g., night shift), a diagnosed sleep disorder, or a chronic medical condition that may impact mood and/or cognition levels, in the judgment of the Investigator.
8. Subject has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg) at visit 1 (day -6).
9. Subject has an active infection or signs/symptoms of an infection. Test visits will be re-scheduled to allow subject to be symptom-free from any type of systemic infection for at least 5 d.
10. Subject has a known allergy or sensitivity to any ingredients in the study products.
11. Subject has used recreational drugs or prescription medications with potential to influence mood, anxiety, cognitive function, and/or modulate the autonomic nervous system (including narcotic (opioid) pain medications) within 4 weeks of visit 1 (day -6).
12. Subject has used nicotine withdrawal/replacement therapy within 6 months of visit 1 (day -6).
13. Subject has used over-the-counter medications, supplements, and/or products, which may influence mood, anxiety, and/or cognitive function within 2 weeks of visit 1 (day -6).
14. Subject has a history of cancer within 5 years prior to visit 1 (day -6), except for non-melanoma skin cancer.
15. Subject is a female, who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded in the source documentation.
16. Subject has a current or recent history (past 12 months of visit 1, day -6) or strong potential for drug or alcohol abuse. Alcohol abuse will be defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1.5 oz hard liquor).
17. Subject has been exposed to any non-registered drug product within 30 d prior to visit 1 (day -6).
18. Individual has a condition the Investigator believes would interfere with his/her ability to provide informed consent, comply with the study protocol, or which might confound the interpretation of the study results, or put the subject at undue risk.

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Mean STAI-Part 1 post-dose score (collected as part of the test battery at the t = 90 and 180 min timepoints) at the end (day 7) of each of the two treatment conditions. | Day 7

SECONDARY OUTCOMES:
Total area under the curve (AUC) for salivary cortisol from 90 to 150 min and 180 to 240 min at the end (day 7) of each of the two treatment conditions | Day 7
Bond-Lader post-dose VAS scores (collected as part of the test battery at the t = 90 and 180 min timepoints) at the end (day 7) of each of the two treatment conditions. | Day 7
Cognitive function post-dose test scores (collected as part of the test battery at the t = 90 and 180 min timepoints) at the end (day 7) of each of the two treatment conditions. | Day 7

OTHER OUTCOMES:
STAI-Part 1 mean and individual timepoint post-dose scores (collected as part of the test battery at the t = 90 and 180 min timepoints) at the start (day 1) of each of the two treatment conditions. | Day 1
Total area under the curve (AUC) for salivary cortisol from 90 to 150 min and 180 to 240 min at the start (day 1) of each of the two treatment conditions. | Day 1
Bond-Lader post-dose VAS scores (collected as part of the test battery at the t = 90 and 180 min timepoints) at the start (day 1) of each of the two treatment conditions. | Day 1
Cognitive function post-dose test scores (collected as part of the test battery at the t = 90 and 180 min timepoints) at the start (day 1) of each of the two treatment conditions | Day 1
Safety will be assessed by vital signs measured at the beginning and end of the study, as well as AEs reported by subjects at each post-randomization clinic visit. | Entire study period
Exploratory analyses will be completed to assess possible predictors of response. | Day 1 and Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Seth J Baum, MD, Principal Investigator — MB Clinical Research; Kevin C Maki, PhD, Study Director — MB Clinical Research
Locations (1):
- MB Clinical Research, Boca Raton, Florida, United States